CLINICAL TRIAL: NCT06256601
Title: A Clinical Investigation of the Effectiveness of a Calcium Silicate Cement Used in the Treatment of Deep Lesions
Brief Title: Clinical Investigation of Effectiveness of a Calcium Silicate Cement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Betul Kesim, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-23024
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Deep Caries; Dentin Caries
Keywords: deep dentin caries; calcium silicate; calcium hydroxide; selective caries removal; randomized clinical trial

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Theracal (calcium silicate) (Experimental): TheraCal LC is a light-cured resin-modified calcium silicate pulp protectant/liner designed to perform as a barrier and to protect the dental pulpal complex. It contains; resin bis-phenyl glycidyl methacrylate (BisGMA) & polyethylene glycol dimethacrylate (PEGD), modified calcium silicated with CaO, calcium silicate particles (type III Portland cement), Sr glass, fumed silica, barium sulphate, barium zirconate.
  After caries removal, TheraCal is applied directly to the cavity floor in incremental layers. The layer is not to exceed 1 mm in depth. Each layer polymerized for 20 seconds.
  Interventions: Device: Theracal (calcium silicate)
- Dycal (calcium hydroxide) (Active Comparator): Dycal,Calcium Hydroxide Liner is a two-component, rigid-setting, self-curing material designed for use in direct and indirect pulp capping and as a protective liner under dental adhesives, varnishes, filling materials, cements, and other base materials. It will not inhibit the polymerization of acrylic and composite restorations. Dycal, a two-paste system made of a base paste (1,3-butylene glycol disalicylate, zinc oxide, calcium phosphate, calcium tungstate, iron oxide pigments) and a catalyst paste (calcium hydroxide, N-ethyl-o/p-toluene sulphonamide, zinc oxide, titanium oxide, zinc stearate, iron oxide pigments) is prepared following the manufacturer's instructions by mixing equal amounts of catalyst paste and base paste.
  After caries removal, Dycal is applied directly to the cavity floor, material thickness should be approximately 0.8mm-1mm. The mixed material will set in approximately 2-3 minutes.
  Interventions: Device: Dycal (calcium hydroxide)

INTERVENTIONS:
Device: Theracal (calcium silicate) — selective removal to soft dentin, restorations with calcium silicate
  Arms: Theracal (calcium silicate)
Device: Dycal (calcium hydroxide) — selective removal to soft dentin, restoration with calcium hydroxide
  Arms: Dycal (calcium hydroxide)

SUMMARY:
The aim of this clinical study is to investigate the clinical performance of a calcium silicate used in the treatment of deep caries lesions. Individuals participating in the research will be selected from patients with at least one deep dentin caries (D3) who apply to the Restorative Dentistry Clinic of Hacettepe University Faculty of Dentistry. The age range will be range 18-45.

The teeth to be restored will be evaluated clinically and radiographically. A rubber dam will be used during the treatment. After the removal of enamel, carious tissue at the lateral walls of cavities will be removed to hard dentin using round and single-use round steel burs operating at low speed in all groups. A reasonable amount of soft carious tissue will be left over the pulp.

In test (Calcium silicate) and control(calcium hydroxide) groups, after caries removal, respective material will be applied on the pulpal floor. Then, materials will be sealed by resin-modified glass ionomer cement and permanent restoration will be performed. Evaluation will be conducted after 6, 12, and 18 months.

DETAILED DESCRIPTION:
This clinical study aims to investigate the 18-month clinical performance of calcium silicate and calcium hydroxide materials used in the treatment of deep caries lesions.

Material and Methods: Eighty patients who applied to the Restorative Dentistry Clinic of Hacettepe University Faculty of Dentistry, aged between 18-45 years, will be recruited for the study. Patients to be included must have at least one deep dentin caries (D3). For standardization purposes, one researcher will carry out the interventional procedures. Before interventions, any attachments on the teeth will be removed using pumice and polishing rubbers. Restorations will be carried out under rubber dam isolation (OptraDam, Liechtenstein). If the patient experiences any pain, anesthesia will be applied. Dentinal carious lesions will be accessed by the removal of surrounding unsupported enamel with a round diamond bur at high speed under water cooling. Carious tissue in the pulpal aspect of the cavity will be excavated by hand instruments to soft dentin. Only disorganized dentine will be removed. A reasonable amount of soft carious tissue will be left over the pulp. The procedure will be carried out considering the risk of exposing the pulp tissue. In the test group a Calcium silicate, (TheraCal LC, Bisco, Schaumburg, IL, USA), and in the control group a calcium hydroxide (Dycal, Dentsply, Caulk, Milford, DE, USA) materials will be applied to the pulpal floor following the instructions of the manufacturer. Then, these materials in both groups will be sealed by resin-modified glass ionomer cement (SDI, Bayswater, Australia).

Selective etching with 37% phosphoric acid (Total Etch-Ivoclar/Vivadent, Liechtenstein) will be applied for 10 s in enamel. Cavities will be rinsed for 10 s, and adhesive material (G-Premio-bond, GC Europe, Leuven, Belgium) will be applied with a micro brush in cavity walls with rubbing for 20 s. After gentle air drying for approximately 5 s, a 1200 W/cm2 intensity LED light device) will be used for 10 s light curing. For the restoration of Class II cavities, a sectional matrix (Palodent V3, Dentsply Sirona, York/Pennsylvania, USA) will be placed. Then, permanent restoration with a posterior composite resin (Gradia Direct Posterior, GC, GC Coop., Tokyo, Japan) will be carried out at the same session. Evaluations will be conducted by two independent researchers after 6, 12, and 18 months according to FDI criteria.

ELIGIBILITY:
Inclusion Criteria:

* The age of the patient should be ranged between 18-45.
* The score of the caries lesion should be D3.
* Absence of a history of spontaneous pain in the teeth to be included.
* Absence of periapical pathology
* No displacement or mobility of the teeth.
* Caries should not have reached the pulp tissue, and there should be no root fractures.
* Restorable by direct restoration and functional

Exclusion Criteria:

* Poor oral hygiene of the participant.
* Parafunctional habits such as teeth clenching or grinding.
* Caries extending to the underneath of gingival margin
* Severe periodontal pathology
* Previous restored teeth
* Teeth undergoing orthodontic treatment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Fracture of restorative material and retention | From Baseline to 12 Month
  Observers evaluated the restorations was performed using FDI criteria regarding fracture of restorative material and retention. Fracture of restorative material and retention was evaluated by 2 independent clinicians. Visual inspection with a mirror was performed. Scores; 1: Restoration retained, no fractures, cracks or chipping 2: Small hairline crack 3: Two or more or larger hairline cracks and/or chipping (not affecting the marginal integrity or proximal contact) 4: Chipping fractures affect marginal quality and/or proximal contacts; bulk fractures with or without partial loss of (<1/2 of the restoration) 5: (Partial or complete) loss of the restoration
Postoperative sensitivity and tooth vitality | From Baseline to 12 Month
  Observers evaluated the restorations was performed using FDI criteria regarding postoperative sensitivity and tooth vitality. Postoperative sensitivity and tooth vitality was evaluated by 2 independent clinicians. Scores; 1: No hypersensitivity, normal vitality 2: Low hypersensitivity for a limited period of time, normal vitality 3: Premature/slightly more intense or delayed/weak hypersensitivity. No subjective complaints 4:Premature/very intense or extremely delayed/weak hypersensitivity with subjective complaints. Or negative sensitivity 5: Very intense, acute pulpitis or non vital tooth. Removal of restoration with or without immediate root canal treatment is required or the tooth must be extracted
Recurrence of initial pathology (secondary caries) | From Baseline to 12 Month
  Observers evaluated the restorations was performed using FDI criteria regarding recurrence of initial pathology (secondary caries). Recurrence of initial pathology (secondary caries) was evaluated by 2 independent clinicians. Visual inspection with a mirror was performed. Scores; 1: No secondary or primary caries 2: Very small, localized demineralization area 3: Larger areas of demineralisation, preventive measures necessary (dentine not exposed) 4: Caries with cavitation 5: Deep secondary caries or exposed dentine that is not accessible for repair
Tooth cracks and fractures | From Baseline to 12 Month
  Observers evaluated the restorations was performed using FDI criteria regarding tooth cracks and fractures. Tooth cracks and fractures was evaluated by 2 independent clinicians. Visual inspection with a mirror was performed. Scores; 1: Complete integrity 2: Minor marginal crack or a hairline crack which cannot be probed. The patient has no clinical symptoms 3: Enamel split or crack <250 μm. No adverse effects 4: Major enamel split (gap >250 μm or dentine/base exposed. Or crack>250 μm (explorer penetrates) 5: Cusp or tooth fracture
Localised reactions of soft tissue | [Time Frame: From Baseline to 12 Month]
  Observers evaluated the restorations was performed using FDI criteria regarding localised reactions of soft tissue. Localised reactions of soft tissue in direct contact with the restoration was evaluated by 2 independent clinicians. Scores; 1: Healthy mucosa adjacent to restoration 2: Healthy after minor removal of mechanical irritations (sharp edges etc.) 3: Alteration of mucosa but no suspicion of causal relationship with filling material 4: Suspected mild allergic, lichenoid or toxicological reaction 5: Suspected severe allergic, lichenoid or toxicological reaction
Oral and somatic/ psychiatric symptoms | [Time Frame: From Baseline to 12 Month]
  Observers evaluated the restorations was performed using FDI criteria regarding oral and somatic/ psychiatric symptoms. Oral and somatic/ psychiatric symptoms in direct contact with the restoration was evaluated by 2 independent clinicians. Scores; 1: No symptoms of adverse effects 2: Short-term minor transient symptoms 3: Minor oral and/or general symptoms of malaise 4: Persistent oral/general symptoms, recurrent symptoms 5: Acute/severe oral/general symptoms requires immediate replacement

CONTACTS AND LOCATIONS:
Overall Officials: Arlin Serpuhi Kiremitci, Prof., Study Director — Hacettepe University; Uzay Koç Vural, Assoc. Prof., Principal Investigator — Hacettepe University; Betül Kesim, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Schwendicke F, Walsh T, Lamont T, Al-Yaseen W, Bjorndal L, Clarkson JE, Fontana M, Gomez Rossi J, Gostemeyer G, Levey C, Muller A, Ricketts D, Robertson M, Santamaria RM, Innes NP. Interventions for treating cavitated or dentine carious lesions. Cochrane Database Syst Rev. 2021 Jul 19;7(7):CD013039. doi: 10.1002/14651858.CD013039.pub2. PMID 34280957
- [Background] Figundio N, Lopes P, Tedesco TK, Fernandes JCH, Fernandes GVO, Mello-Moura ACV. Deep Carious Lesions Management with Stepwise, Selective, or Non-Selective Removal in Permanent Dentition: A Systematic Review of Randomized Clinical Trials. Healthcare (Basel). 2023 Aug 18;11(16):2338. doi: 10.3390/healthcare11162338. PMID 37628535
- [Background] Schwendicke, F., in Management of Deep Carious Lesions. 2018, Springer Nature: Gewerbestrasse.
- [Background] Innes NP, Frencken JE, Bjorndal L, Maltz M, Manton DJ, Ricketts D, Van Landuyt K, Banerjee A, Campus G, Domejean S, Fontana M, Leal S, Lo E, Machiulskiene V, Schulte A, Splieth C, Zandona A, Schwendicke F. Managing Carious Lesions: Consensus Recommendations on Terminology. Adv Dent Res. 2016 May;28(2):49-57. doi: 10.1177/0022034516639276. PMID 27099357
- [Background] Barros MMAF, De Queiroz Rodrigues MI, Muniz FWMG, Rodrigues LKA. Selective, stepwise, or nonselective removal of carious tissue: which technique offers lower risk for the treatment of dental caries in permanent teeth? A systematic review and meta-analysis. Clin Oral Investig. 2020 Feb;24(2):521-532. doi: 10.1007/s00784-019-03114-5. Epub 2019 Nov 26. PMID 31773371
- [Background] Kunert M, Lukomska-Szymanska M. Bio-Inductive Materials in Direct and Indirect Pulp Capping-A Review Article. Materials (Basel). 2020 Mar 7;13(5):1204. doi: 10.3390/ma13051204. PMID 32155997
- [Background] Schmidt J, Buenger L, Krohn S, Kallies R, Zeller K, Schneider H, Ziebolz D, Berg T, Haak R. Effect of a bioactive cement on the microbial community in carious dentin after selective caries removal - An in-vivo study. J Dent. 2020 Jan;92:103264. doi: 10.1016/j.jdent.2019.103264. Epub 2019 Dec 13. PMID 31843419
- [Background] Koc Vural U, Kiremitci A, Gokalp S. Which is the most effective biomaterial in indirect pulp capping? 4- year comparative randomized clinical trial. Eur Oral Res. 2022 Jan 1;56(1):35-41. doi: 10.26650/eor.2022895748. PMID 35478709
- [Background] Edwards D, Stone S, Bailey O, Tomson P. Preserving pulp vitality: part one - strategies for managing deep caries in permanent teeth. Br Dent J. 2021 Jan;230(2):77-82. doi: 10.1038/s41415-020-2590-7. Epub 2021 Jan 22. PMID 33483661
- [Background] Jurasic MM, Gillespie S, Sorbara P, Clarkson J, Ramsay C, Nyongesa D, McEdward D, Gilbert GH, Vollmer WM; National Dental PBRN Collaborative Group. Deep caries removal strategies: Findings from The National Dental Practice-Based Research Network. J Am Dent Assoc. 2022 Nov;153(11):1078-1088.e7. doi: 10.1016/j.adaj.2022.08.005. Epub 2022 Sep 26. PMID 36175201